CLINICAL TRIAL: NCT07377487
Title: A Prospective Single-arm Study of BSJ019T in Japanese Patients With Unresectable Hepatic Malignancy Who Have Failed or Are Not Eligible for Standard Treatment
Brief Title: TheraSphere Japan Pre-Market Study
Acronym: INDIGO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2486
Record Dates: First submitted 2025-09-24; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Liver Neoplasms
Keywords: Carcinoma; Carcinoma, Hepatocellular; Neoplasms; Digestive System Neoplasms; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms by Site; Digestive System Diseases; Liver Diseases; Neoplasm Metastasis; Colorectal Neoplasms; Colonic Diseases; Carcinoma, Neuroendocrine; Neuroendocrine Tumors
MeSH Terms: conditions — Liver Neoplasms; Carcinoma; Carcinoma, Hepatocellular; Neoplasms; Digestive System Neoplasms; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms by Site; Digestive System Diseases; Liver Diseases; Neoplasm Metastasis; Colorectal Neoplasms; Colonic Diseases; Carcinoma, Neuroendocrine; Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TheraSphere (Experimental)
  Interventions: Device: TheraSphere Y-90 glass microsphere

INTERVENTIONS:
Device: TheraSphere Y-90 glass microsphere — TheraSphere Y-90 glass microsphere therapy administered through the hepatic artery at index procedure.

SUMMARY:
To investigate the safety and effectiveness of BSJ019T in Japanese patients with primary or secondary liver who are not candidate for standard treatment.

ELIGIBILITY:
Inclusion Criteria:

[Inclusion criteria based on the clinical evaluation]

1. Patient aged >18 years at time of consent
2. Patient is able and willing to participate in the study and has provided written informed consent
3. Patient who is determined to have failed or not be eligible for standard treatment by the multidisciplinary board
4. Primary or secondary liver cancer (by histology or imaging)
5. Measurable disease defined as at least one uni-dimensional measurable liver lesion by CT/MRI (according to RECIST 1.1)
6. Liver dominant disease (patient prognosis is driven by liver tumor)
7. Tumor replacement <50% of total liver volume based on visual estimation by the investigator
8. Expected life expectancy ≥ 3 months or more from the index procedure
9. ECOG Performance Status score of 0 or 1
10. Negative pregnancy test in women of child-bearing potential
11. Adequate contraception for the patient and his/her sexual partner when applicable.
12. Adequate liver function, as defined by:

    * Child Pugh A or to B7 (HCC)
    * Must have bilirubin ≤ 2 mg/dL
    * ALT and AST must be <5 x ULN
    * Albumin ≥3.0 g/dL
13. Adequate renal function, as defined by:

    • Serum creatinine must be ≤1.5 x ULN
14. Adequate hematological function, as defined by:

    * Neutrophil count > 1200 /mm3
    * hemoglobin ≥85 mg/L
    * platelet count >50 x 109/L
    * INR must be <2.0 or >50% prothrombin activity

    [Inclusion Criteria based on the imaging evaluation]
15. After 99mTc MAA administration, in SPECT/CT imaging, good PVT targeting and uptake of 99mTc MAA, if present
16. Future liver remnant volume (FLRV) >30% of whole liver volume. FRLV is the volume of liver not planned to be treated with TheraSphere and free of tumor

Exclusion Criteria:

[Exclusion Criteria based on the clinical evaluation]

1. Vp4 according to the Liver Cancer Study Group of Japan (LCSGJ) portal vein tumor thrombosis classification1
2. History of severe allergy or intolerance to contrast agents, narcotics sedatives or atropine that cannot be managed medically.
3. Contraindications to angiography and selective visceral catheterization
4. Received any prior external beam radiation treatment to the liver
5. Received any prior yttrium-90 microsphere treatment to the liver
6. Received previous peptide receptor radionuclide therapy (PRRT)
7. Plan to start systemic anticancer treatment in the next 3 month after the index procedure.
8. Presence of ongoing adverse event due to prior therapy as judged by the principal investigator or sub-investigator to affect the safety evaluation of the study device.
9. Evidence of pulmonary insufficiency or clinically evident chronic obstructive pulmonary disease
10. Undergone any intervention for, or compromise of, the Ampulla of Vater within that last 3 months or patient with biliodigestive anastomosis.
11. Presence of ascites, clinical or radiological, "trace" of ascites is acceptable.
12. Presence of Hepatic encephalopathy (Grade ≥2)
13. Previous liver function decompensation within the last 6 months (ascites, encephalopathy, jaundice)
14. Patient with infiltrative disease presentation (not suitable for repeated measurement)
15. Patients who are pregnant or breast-feeding and does not want to stop.
16. Have any disease or condition that would preclude the safe use of BSJ019T, including concurrent dialysis treatment, or unresolved serious infections
17. Participating in concurrent clinical studies or interventional clinical studies
18. Any condition where the Investigator feels the patient would not be able to participate/finish the study
19. Previous gastrointestinal bleeding related to portal hypertension within the last 3 months (preventive treatment is acceptable)

    [Exclusion Criteria based on the imaging evaluation]
20. Dose to the lung > 30Gy for a single treatment or cumulative >50 Gy
21. Evidence of any off-target extrahepatic and liver deposition on 99mTc-MAA that cannot be corrected using angiographic techniques
22. Cone Beam CT (CBCT) or 99mTc-MAA hepatic arterial perfusion scintigraphy shows poor tumor perfusion and/or poor tumor targeting that would lead to a dose that does not meet the liver dosing criteria as specify in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2026-01-22 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Rate of hepatic disease control (DCR = complete response [CR], partial response [PR] or stable disease [SD]) at 3 months using the localized RECIST 1.1 criteria. | 3-months post index procedure

SECONDARY OUTCOMES:
Rate of objective response (ORR = complete response [CR] or partial response [PR]) at 3 months using the localized RECIST 1.1 criteria and localized mRECIST | 3-months post index procedure
Rate of hepatic disease control (DCR) and objective response (ORR) at 6 months using localized RECIST 1.1 and localized mRECIST criteria | 6-months post index procedure
Best response using localized RECIST 1.1 and localized mRECIST criteria. | Through 6-months post index procedure
Proportion of patient receiving concomitant and post BSJ019T treatment, including subsequent local and systemic anticancer treatment, surgery, intervention and best supportive care. | Through 6-months post index procedure
Safety assessment: rate of treatment emergent adverse events (TEAEs) of any grade, rate of grade 3 or above TEAEs, rate of SAEs of any causality and rate of SAEs related to treatment with TheraSphere. | Through 6-months post index procedure
  All AEs will be evaluated using the standardized grading criteria (National Cancer Institute- Common Terminology Criteria for Adverse Events- Version 5.0 (NCI-CTCAE v 5.0))
Technical success in delivering the Y-90 microspheres | During the index procedure
  Technical success is determined successful if residual waste is ≦2% with optimal tumor targeting and extrahepatic deposition is not seen on post treatment imaging, and the success rate of entire of the subjects will be summarized.
Health-related quality of life (HRQoL) using EQ-5D questionnaires at regular intervals | Baseline, 1-, 3- and 6-months post treatment
Health-related quality of life (HRQoL) using FACT-G questionnaires at regular intervals | Baseline, 1-, 3- and 6-months post treatment
Overall survival | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Koichiro Yamakado, MD, PhD, Principal Investigator — Hyogo Medical University
Locations (4):
- Japan (4):
  - Hyogo College of Medicine Hospital, Nishinomiya, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kindai University Hospital, Sayama, Osaka
  - National Cancer Center Hospital, Chuo Ku, Tokyo

IPD SHARING:
Plan to Share IPD: No